CLINICAL TRIAL: NCT03560557
Title: Optimization of PK/PD Target Attainment for Meropenem in Critically Ill Patients With Sepsis
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Matthias Gijsen, PharmD, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: ML8459
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Critical Illness; Pharmacokinetics
Keywords: Pharmacokinetics; Meropenem; Critical illness; Capillary leak; Augmented renal clearance
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, urine, bronchoalveolar lavage fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
WP1.1. PK/PD target attainment: Plasma exposure, Excretion via urine & ELF exposure; WP1.2. Predictive dosing algorithm; WP1.3. ECMO subset

DETAILED DESCRIPTION:
First, the investigators will document exposure to meropenem in plasma and epithelial lining fluid. Moreover excretion in urine will be documented.

Second, the investigators will try to identify risk factors for not attaining PK/PD target. Based on significant predictors for target non attainment a predictive dosing algorithm will be constructed.

Finally in a small subset of ECMO patients PK exposure will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis or septic shock
* Admitted to an ICU ward
* Treated with meropenem

Exclusion Criteria:

* eGFR(CKD-EPI) < 70ml/min/1.73m²
* Renal replacement therapy
* Pregnancy
* DNR code 1-3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with sepsis and receiving meropenem
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Risk factors for target non attainment | on day of sampling
  risk factors will be assessed by comparing patients who attain target vs. those who don't

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Spriet, PharmD PhD, Study Director — UZ Leuven

IPD SHARING:
Plan to Share IPD: Undecided
To be discussed

REFERENCES:
- [Derived] Gijsen M, Elkayal O, Annaert P, Van Daele R, Meersseman P, Debaveye Y, Wauters J, Dreesen E, Spriet I. Meropenem Target Attainment and Population Pharmacokinetics in Critically Ill Septic Patients with Preserved or Increased Renal Function. Infect Drug Resist. 2022 Jan 8;15:53-62. doi: 10.2147/IDR.S343264. eCollection 2022. PMID 35035223